CLINICAL TRIAL: NCT00479206
Title: Artemisinin Resistance in Cambodia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Global Emerging Infections Surveillance and Response System (U.S. Federal Agency); Armed Forces Research Institute of Medical Sciences, Thailand (Other Government); National Center for Parasitology, Entomology and Malaria Control (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WRAIR #1296; HSRRB A-13922
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Last update posted 2008-04-30 (Estimated); Status verified 2008-04

CONDITIONS: Malaria, Falciparum
Keywords: artesuante; falciparum malaria; Cambodia; Artemisinin resistance
MeSH Terms: conditions — Malaria, Falciparum | interventions — Artesunate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Artesunate

SUMMARY:
The principal aim of this project is to investigate reports of developing artemisinin resistance in Cambodia using an integrated in vivo - in vitro approach to examine recent alarming reports of treatment failures with advanced combination therapies along the Thai-Cambodian border, which could have major impact on the malaria situation in the affected areas as well as the rest of the malaria-endemic world.

DETAILED DESCRIPTION:
A total number of 90 volunteers with acute uncomplicated falciparum malaria will be randomly assigned to be treated with either artesunate monotherapy for 7 days or the combination of quinine and tetracycline over 7 days (following the 2nd line national treatment guideline of the national malaria control program) at a ratio of 2:1. The study design will be based on the WHO recommendations for the 'Assessment and Monitoring of Antimalarial Drug Efficacy for the Treatment of Uncomplicated Falciparum Malaria' (WHO, 2003). Study participants will be otherwise healthy malaria patients (adult men and non-pregnant women aged 18 to 65 years) with uncomplicated falciparum malaria recruited in Battambong Province, Cambodia.

The artesunate will be administered orally (a single dose of 200 mg per day) over a total duration of 7 days (Directly Observed Therapy). Quinine (30 mg/kg/day) plus tetracycline (25 mg/kg/day) will also be administered over 7 days in split dose every 8 hours following the national treatment guidelines of Cambodia.

Patients will be admitted to the hospital for the duration of study drug administration or until all signs and symptoms of malaria have disappeared, whichever comes first. Thereafter until Day 21 patients have to remain in a malaria-free environment (such as Sampov Luon or Ta Sanh) either in the hospital or in a living facility provided at the study site where the patients will be supervised by study personnel. After Day 21 they will be followed as outpatients until Day 28 with a scheduled follow-up visit on Day 28.

In vitro drug sensitivity assays will be performed from samples on inclusion and in case of recrudescence. Drug levels will be measured in the artesunate arm on the first and last day of therapy.

Primary clinical outcome is cure (Adequate Clinical and Parasitological Response - ACPR) on Day 28. Secondary outcome measures are time until parasite, fever, and gametocyte clearance (PCT, FCT, and GCT). Parasite genotyping will be used to distinguish recrudescences from reinfections by PCR. Subjects will be monitored for clinical adverse events throughout the study duration.

Blood will be drawn on the day of admission (before initiating therapy) for in vitro drug sensitivity testing and for PCR (markers of drug resistance and to distinguish recrudescence from reinfection by genotyping). Malaria smears will be prepared up to 4 times a day until parasite clearance and on Days 7, 14, 21, and 28 or whenever symptoms consistent with malaria appear. Plasma samples for determining drug levels will be obtained on the first and last day of therapy. Over the entire study, up to approximately 64 ml of blood may be drawn by venipuncture. Study participation for each individual will be 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Acute symptomatic falciparum malaria infection as determined by malaria smear with a parasite density of 100 to 100,000 asexual parasites/uL as determined on the screening smear with fever (defined as >=37.5ºC), or reported history of fever within the last 48 hours.
* Age: 18-65 years old
* Males or females. All females are required to have a negative human chorionic gonadotropin (hCG) pregnancy test (urine). All females of childbearing potential (not surgically sterile, or less than two years menopausal) are required to use an acceptable method of contraception, such as implant, injectable, oral contraceptive(s) with additional barrier contraception, intrauterine device, sexual abstinence, or vasectomized partner, throughout the study
* Written informed consent obtained
* Willing to stay under close medical supervision for the study duration of 28 days
* Otherwise healthy outpatients

Exclusion Criteria:

* Pregnant women, nursing mothers, or women of childbearing potential who do not use an acceptable method of contraception (as described in Inclusion Criteria, #3)
* Mixed malaria infection on admission by malaria smear
* A previous history of intolerance or hypersensitivity to the study drugs artesunate, quinine, or tetracycline or to drugs with similar chemical structures (quinidine, any artemisinin derivative, and tetracyclines)
* Malaria drug therapy administered in the past 30 days by history
* Previous participation in this trial, or participation in any other studies involving investigational or marketed products, concomitantly or within 30 days prior to entry in the study
* History of significant cardiovascular, liver or renal functional abnormality or any other clinically significant illness, which in the opinion of the investigator would place them at increased risk.
* Symptoms of severe vomiting (no food or inability to take food during the previous 8 hours).
* Signs or symptoms of severe malaria (as defined by WHO 2003)
* Unable and/or unlikely to comprehend and/or follow the protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-10; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Primary clinical outcome is cure (Adequate Clinical and Parasitological Response - ACPR as defined by WHO criteria) on Day 28.

SECONDARY OUTCOMES:
Secondary outcome measures are time until parasite, fever, and gametocyte clearance (PCT, FCT, and GCT).

CONTACTS AND LOCATIONS:
Overall Officials: Harald Noedl, MD, MCTM, PhD, Study Director — USAMC-AFRIMS
Locations (1):
- Tasanh Health Center, Tasanh, Battambang, Cambodia

REFERENCES:
- [Derived] Noedl H, Se Y, Sriwichai S, Schaecher K, Teja-Isavadharm P, Smith B, Rutvisuttinunt W, Bethell D, Surasri S, Fukuda MM, Socheat D, Chan Thap L. Artemisinin resistance in Cambodia: a clinical trial designed to address an emerging problem in Southeast Asia. Clin Infect Dis. 2010 Dec 1;51(11):e82-9. doi: 10.1086/657120. Epub 2010 Oct 28. PMID 21028985